CLINICAL TRIAL: NCT04182217
Title: Descriptive and Correlational Study of the Epidemiological, Clinical and Etiological Characteristics of Peritonitis in the Surgical Department of the State University Hospital of Haiti During the Period From January 2013 to December 2018
Brief Title: Descriptive and Correlational Study of Peritonitis in Haiti.
Status: Completed | Type: Observational
Sponsor: Universite d'Etat d'Haiti (Other)
Responsible Party: Principal Investigator, JEAN PAUL Axler, Medical Student, Universite d'Etat d'Haiti
Other Study IDs: 01
Record Dates: First submitted 2019-11-23; First posted 2019-12-02 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Epidemiological description — Description of the characteristics of Peritonitis in Haiti

SUMMARY:
The primary objective:

To study the prevalence, etiology, and factors associated with the severity of peritonitis and its complications in the surgery department of the State University Hospital of Haiti.

Secondary objectives:

* Identify epidemiological characteristics.
* Describe the main etiologies encountered in the service
* Measure the time required for treatment and its consequences on the evolution of peritonitis.

DETAILED DESCRIPTION:
Generalized secondary peritonitis is one of the most common emergencies encountered in surgical departments . It is a major surgical condition with a mortality of up to 20% and classified as the third most common cause of surgical abdomens after appendicitis and intestinal obstruction . Delays in surgical management are conditions that increase mortality. While early prognostic assessment of peritonitis is essential for the objective classification of the severity of the disease, the late presentation of the majority of patients to health facilities affects this situation, further complicating effective management and promoting the occurrence of complications . It has been observed that classifying the severity of peritonitis has a major contribution to decision-making and improves management. Thus, many scoring systems have been designed and successfully used to assess the severity of acute peritonitis, including: Acute physiology and chronic health evaluation (APACHE) II score, Simplified acute physiology score (SAPS), Sepsis severity score (SSS), Ranson score, Imrite score, Mannheim peritonitis index (MPI) 6. The Mannheim Peritonitis Index (MPI) is a specific score, which is highly accurate and allows clinical parameters to be easily manipulated, allowing the individual prognosis of patients with peritonitis to be predicted . In Haiti, few studies on surgical pathologies are available. And with regard to peritonitis, only two thesis works have been listed on the subject, including one carried out at the Justinian University Hospital of Cap-Haitian on 176 patients by Dr. Jacques Julmice, who presents the main etiologies of peritonitis over a 5-year period. And the other one carried out at the Albert Schweizer Hospital by Dr. Moise Aristide, still on the etiological factors of peritonitis. These two studies are carried out outside the country's metropolitan region (the most populated region) and that they only explored the different etiologies without taking into account the time required for treatment and the gravity factors of peritonitis. Therefore, our study aims to explore the demographic, clinical and etiological factors of peritonitis in the main referral hospital in the metropolitan region of the country, as well as the time required for treatment and its relationship with the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

Patients whose peritonitis diagnosis was made and operated on in the department during the period.

Patient whose record is identified (with age, sex) with at least the clinical and etiological diagnosis identified in the operating protocol.

Exclusion Criteria:

Patients with incomplete records.

Cases of post-operative peritonitis.

Patient under 10 years of age

Ages: 11 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of all patients diagnosed, hospitalized and operated on in the peritonitis ward during the study period.
  Sampling is probabilistic, simple random sampling. To estimate the sample size, we considered the peritonitis prevalence of an African study on the particularity of peritonitis in tropical environments, an environment that reflects our reality in ecological, demographic and epidemiological terms, namely 19% . The standard error rate chosen was 5%. This allows us to estimate our sample at 88 with a confidence interval of 97%. Given the possibility of finding missing files at the State University Hospital of Haïti, our sample was adjusted to 20% (standard non-response rate).
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sterman Toussaint, MD, Study Director — Universite d'Etat d'Haiti
Locations (1):
- Axler JEAN PAUL, Port-au-Prince, Ouest, Haiti

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Population: The study population is composed of all patients diagnosed, hospitalizedand operated on in the peritonitis ward during the study period. Samplingis probabilistic, simple random sampling. To estimate the sample size, weconsidered the peritonitis prevalence of an African study on the particularityof peritonitis in tropical environments, an environment that reflects our realityin ecological, demographic and epidemiological terms, namely 19% . Thestandard error rate chosen was 5%. This allows us to estimate our sample at88 with a confidence interval of 97%. Given the possibility of finding missingfiles at the State University Hospital of Haïti, our sample was adjusted to 20%(standard non-response rate).
Period: Overall Study
Arm/Group | Population
Started | 91
Completed | 91
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Sampling is probabilistic, simple random sampling. To estimate the sample size, weconsidered the peritonitis prevalence of 19% . The standard error rate chosen was 5%. This allows us to estimate our sample at 88 with a confidence interval of 97%. our sample was adjusted to 20%.15 were excluded What makes 91 as the final sample.
Arm/Group | Population
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants] — Population: To estimate the sample size, weconsidered the peritonitis prevalence of 19% . The standard error rate chosen was 5%. This allows us to estimate our sample at 88 with a confidence interval of 97%. our sample was adjusted to 20%.15 were excluded What makes 91 as the final sample.
  Participants
    <=18 years | 30
    Between 18 and 65 years | 58
    >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.29 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Haiti | 91

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Heart rate number of beats/min reported in the file entry for each patients
Time Frame: immediately after admission, up to 30 minutes
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Population
Number analyzed (Participants) | 86
Beats/min | 108.18 (19.66)

2. Primary Outcome: Respiratory Rate
Description: Respiratory rate number of cycle/min reported in the file of entry
Time Frame: immediately after admission, up to 30 minutes
Population: For the other (11) patients we did not find any data relating to the respiratory rate.
Measure: Mean (Standard Deviation); unit: Cycle/min
Arm/Group | Population
Number analyzed (Participants) | 80
Cycle/min | 28.58 (8.51)

3. Primary Outcome: Temperature
Description: Temperature in celsius reported in the file of entry
Time Frame: immediately after admission, up to 30 minutes
Population: For the other (6) patients we did not find any data relating to the temperature
Measure: Mean (Standard Deviation); unit: Celcius
Arm/Group | Population
Number analyzed (Participants) | 85
Celcius | 37.52 (1.1)

4. Primary Outcome: Blood Pressure
Description: Systolic Blood pressure in mmHg reported in the file of entry
Time Frame: immediately after admission, up to 30 minutes
Population: For the other (21) patients we did not find any data relating to the systolic blood pressure.
Measure: Mean (Standard Deviation); unit: Hg mm
Arm/Group | Population
Number analyzed (Participants) | 69
Hg mm | 110.93 (14.86)

5. Primary Outcome: Etiological Diagnosis
Description: final diagnosis retained in the operating protocol
Time Frame: immediately post-surgery
Reporting Status: Not Posted

6. Primary Outcome: Demographic Parameters
Description: Age in years described in the admission file
Time Frame: during admission
Reporting Status: Not Posted

7. Secondary Outcome: Onset of Symptoms
Description: Days before coming at the hospital
Time Frame: immediately after admission
Population: We did not find information in the files on the onset of symptoms for 10 patients
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Population
Number analyzed (Participants) | 81
days | 6.9 (8.1)

8. Secondary Outcome: Delay in Pre-op
Description: the pre-operative time in days which describes the time between the date of the intervention and the date of admission
Time Frame: immediately post-surgery
Population: We did not find information in the files on the delay in pre-op for 1 patient
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Population
Number analyzed (Participants) | 90
days | 3.73 (3.61)

9. Secondary Outcome: Delay in Post-op
Description: the time in days between the date of the intervention and the leaving of the patient at the hospital
Time Frame: immediately after hospitalization
Population: We did not find information in the files on the delay in post-op for 1 patient
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Population
Number analyzed (Participants) | 90
days | 9.19 (10.93)

10. Secondary Outcome: Delay in Hospital
Description: the time in days between the date of admission and the date of leaving the hospital
Time Frame: immediately after hospitalization
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Population
Number analyzed (Participants) | 91
days | 12.82 (11.66)

ADVERSE EVENTS:
Time Frame: 24 hours in post-operation rooms
Description: The adverse events were the cases of post-operative complications recorded during the study.
Arm/Group | Population
All-Cause Mortality (participants affected / at risk) | 3/91
Serious Adverse Events (participants affected / at risk) | 21/91
Other Adverse Events (participants affected / at risk) | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Population (N=91)
Post-operative complications (Surgical and medical procedures) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04182217/Prot_SAP_001.pdf